CLINICAL TRIAL: NCT04514926
Title: Blood Lymphocytes in Asthmatics Treated With Therapeutic Proteins
Acronym: BLAST
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 20-30026; 2P01HL107202-06A1 (NIH)
Record Dates: First submitted 2020-08-12; First posted 2020-08-17 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Asthma; Therapeutic Proteins
Keywords: asthma; therapeutics; therapeutic proteins
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Controls: Participants with no history of asthma or other lung diseases.
- Asthmatics newly prescribed therapeutic proteins: Participants with asthma, have been newly prescribed therapeutic proteins and have yet to start on those therapeutics at the time of enrollment.
- Asthmatics already being treated with therapeutic proteins: Participants with asthma who have already started on therapeutic proteins.

SUMMARY:
This is an observational, clinic-based, single center study of 120 subjects. Participants will be comprised of patients seen in the outpatient faculty practice in ambulatory care at the UCSF Parnassus campus. Study investigators will enroll 20 healthy participants with no history of lung disease, 50 asthmatics who are newly prescribed therapeutic proteins for their asthma, and 50 asthmatics already being treated with therapeutic proteins for their asthma. Participants will be seen at 1 to 3 visits and provide blood samples at each visit.

DETAILED DESCRIPTION:
Asthma is a common disease affecting 5 - 10% of the population. The main underlying pathology is airway inflammation, which in a majority of patients is characterized by upregulation of type 2 cytokines and infiltration of the airway mucosa with type 2 inflammatory cells. Despite incomplete understanding of mechanisms by which these molecules and cells initiate and propagate the inflammatory process, several new therapies have been developed and even approved to target type 2 cytokines like IL-4, IL-5 and IL13 in asthmatics.

While mechanistic understanding lags behind therapeutic advance, the emergence of these new therapeutics and increase use in treatment of asthmatic patients provides a unique opportunity to better understand how these medicines alter inflammation and ameliorate disease activity. The over-arching goal of this project is to advance understanding of how these new therapeutic proteins modulate inflammation in peripheral blood. A better understanding of these mechanisms will allow for tracking of cellular and molecular biomarkers that may inform treatment regimens with these new therapeutics in patients with asthma.

Through this observational, clinic-based, single center study of 120 subjects, investigators will compare blood lymphocytes as well as other molecular biomarkers associated with inflammation in healthy controls, asthmatic patients not on therapeutic proteins and asthmatics treated with therapeutic proteins. Participants will be comprised of patients seen in the outpatient faculty practice in ambulatory care at the UCSF Parnassus campus. Participants will be seen at 1 to 3 visits and provide blood samples at each visit. It is anticipated that this study will help uncover mechanisms of response to these novel therapeutic interventions in asthma.

ELIGIBILITY:
Group 1:

Inclusion Criteria:

* Male or female between the ages of 18 and 80 years at Visit 1 and at least 50% whose age is >40 years (to ensure age balance among groups and anticipating that groups 1 and 2 will be older).
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.
* Able to perform reproducible spirometry according to ATS criteria.

Exclusion Criteria:

* History of asthma or other lung disease.
* History of allergic rhinitis.
* URI within the previous 6 weeks.
* Smoking of tobacco or other recreational inhalants in last month and/or >10 pack-year smoking history.
* Currently pregnant.
* Abnormal spirometry.

Group 2

Inclusion Criteria

* Male or female between the ages of 18 and 80 years at Visit 1
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.
* Able to perform reproducible spirometry according to ATS criteria.
* Asthma requiring treatment with therapeutic proteins but not yet started on treatment.

Exclusion Criteria

* Asthma exacerbation or URI (upper respiratory infection) within the previous 6 weeks.
* Smoking of tobacco or other recreational inhalants in last month and/or >10 pack-year smoking history.
* Currently pregnant.
* Other chronic pulmonary disorders, including cystic fibrosis and chronic obstructive pulmonary disease.
* Use of other therapeutic proteins in the past 6 months.

Group 3

Inclusion Criteria:

* Male or female between the ages of 18 and 80 years at Visit 1
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.
* Able to perform reproducible spirometry according to ATS criteria.
* Asthma already being treated with therapeutic proteins for at least 6 months.

Exclusion Criteria

* Asthma exacerbation or URI within the previous 6 weeks.
* Smoking of tobacco or other recreational inhalants in last month and/or >10 pack-year smoking history.
* Currently pregnant.
* Other chronic pulmonary disorders, including cystic fibrosis and chronic obstructive pulmonary disease.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Asthmatic patients seen in the outpatient chest faculty practice (clinic) at UCSF Parnassus campus.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Number of Lymphocyte | Up to 18 months
  The investigators will compare lymphocyte counts in healthy controls to asthmatics on and off therapeutic proteins.

CONTACTS AND LOCATIONS:
Overall Officials: John V Fahy, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers.

REFERENCES:
- See also: Airway Clinical Research Center website — http://acrc.ucsf.edu